CLINICAL TRIAL: NCT02289456
Title: A Phase II, Single Arm, Open-Label, Multicenter, Safety and Tolerability Trial With Nab-Paclitaxel (ABRAXANE®) Plus Carboplatin Followed by Nab-Paclitaxel Monotherapy as First-Line Treatment for Subjects With Locally Advanced or Metastatic Nonsmall Cell Lung Cancer (NSCLC) and an Eastern Cooperative Oncology Group Performance Status of 2 (ABOUND.PS2)
Brief Title: Phase II Safety and Tolerability Trial With Nab-Paclitaxel Plus Carboplatin Followed by Nab-Paclitaxel for First Line Treatment of NSCLC Subjects With ECOG PS 2
Acronym: AboundPS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-NSCL-004
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Phase II, LOCALLY ADVANCED OR METASTATIC NON SMALL; CELL LUNG CANCER (NSCLC) AND AN; EASTERN COOPERATIVE ONCOLOGY GROUP; PERFORMANCE STATUS OF 2; (ABOUND.PS2); LOCALLY ADVANCED OR METASTATIC NON SMALL; CELL LUNG CANCER (NSCLC) SUBJECTS THAT AE NOT CANDIDATES FOR RADIATION OR CURATIVE SURGERY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-Paclitaxel (Experimental): nab-Paclitaxel 100 mg/m2 intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle
  • Carboplatin AUC = 5 mg*min/mL IV on Day 1 of each 21-day cycle after completion of nab-paclitaxel infusion.
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: nab-Paclitaxel
  Other Names: Abraxane
Drug: Carboplatin
  Other Names: Paraplatin

SUMMARY:
4 cycles of induction treatment with nab-paclitaxel and carboplatin followed by nab-paclitaxel monotherapy for those subjects who are progression free at the end of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* General and Demographics

  1. Age ≥ 18 years of age at the time of signing the Informed Consent Form.
  2. Understand and voluntarily provide written consent to the Informed Consent Form prior to conducting any study related assessments/procedures.
  3. Able to adhere to the study visit schedule and other protocol requirements. Disease Specific
  4. Histologically or cytologically confirmed Stage IIIB or IV Non-Small Cell Lung Cancer.
  5. Radiographically documented measurable disease at study entry per response evaluation criteria in solid tumours ( RECIST) v1.1.
  6. No prior anti-cancer therapy for the treatment of metastatic disease at the time of signing the ICF. Adjuvant treatment is permitted providing cytotoxic chemotherapy was completed 12 months prior to signing the ICF and without disease recurrence.
  7. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3.
  8. Platelets ≥ 100,000 cells/mm3.
  9. Hemoglobin (Hgb) ≥ 9 g/dL.
  10. Aspartate transaminase (AST/serum glutamic oxaloacetic transaminase [SGOT]), alanine transaminase (ALT/serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × upper limit of normal range (ULN) or ≤ 5.0 × ULN if liver metastases.
  11. Total bilirubin ≤ 1.5 × ULN except in cases of Gilbert's disease and liver metastases.
  12. Serum creatinine ≤ 1.5 x ULN, or calculated creatinine clearance ≥ 40 mL/min (if renal impairment is suspected 24-hour urine collection for measurement is required).
  13. Eastern Cooperative Oncology Group Performance Status 2.
  14. Females of childbearing potential [defined as a sexually mature woman who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months)] must:

      1. Have a negative pregnancy test Beta Human Chorionic Gonaditrophin(ß-hCG) as verified by the study doctor within 72 hours prior to starting study therapy.
      2. You must commit to complete abstinence from heterosexual contact, or agree to use medical doctor-approved contraception throughout the study without interruption; while receiving study medication or for a longer period if required by local regulations.

         Male subjects must:
      3. practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 6 months following study drug discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Evidence of active brain metastases, including leptomeningeal involvement (prior evidence of brain metastasis are permitted only if treated and stable and off therapy for at least 21days prior to signing ICF). MRI of the brain (or CT scan w/contrast) is preferred for diagnosis.
  2. History of leptomeningeal disease.
  3. Only evidence of disease is non-measurable.
  4. Pre-existing peripheral neuropathy of Grade 2, 3, or 4 (per Criteria for Adverse Events (CTCAE) v4.0).
  5. Subject has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting investigational product (IP), and/or from whom ≥ 30% of the bone marrow was irradiated. Prior radiation therapy to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.
  6. Venous thromboembolism within 1 month prior to signing ICF.
  7. Current congestive heart failure (New York Heart Association Class II-IV).
  8. History of the following within 6 months prior to first administration of investigational product: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant ECG abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder.
  9. Subject has a known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications.
  10. Subject has an active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
  11. History of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis.
  12. Treatment with any investigational product within 28 days prior to signing the ICF.
  13. History of or suspected allergy to nab-paclitaxel, carboplatin and human albumin or any other platinum-based therapy.
  14. Currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices.
  15. Any other clinically significant medical condition, psychiatric illness, and/or organ dysfunction that will interfere with the administration of the therapy according to this protocol or which, in the views of investigator, preclude combination chemotherapy.
  16. Subject has any other malignancy within 5 years prior to signing the ICF. Exceptions include the following: squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer (Tumor, node and metastasis (TNM) stage of T1a or T1b). All treatment should have been completed 6 months prior to signing ICF.
  17. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
  18. Any medical condition that confounds the ability to interpret data from the study. This includes subjects with known psychiatric disorders.
  19. Pregnant or breast-feeding females.
  20. Subjects with an ECOG PS other than 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lafleur, MD, Study Director — Celgene Corporation
Locations (8):
- United States (8):
  - University Cancer Institute, Boynton Beach, Florida
  - Ochsner Clinic Nephrology, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - University of RochesterJames P. Wilmont Cancer Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the United States (US) and enrolled participants at 7 sites.
Pre-assignment Details: Included participants with confirmed Stage IIIB or IV non-small cell lung cancer and measurable disease at study entry per Response Evaluation Criteria in Solid Tumors Version 1.1 with an Eastern Cooperative Oncology Group Performance Status of 2 and no prior anticancer therapy for the treatment of metastatic disease.
Groups:
- Nab-Paclitaxel and Carboplatin: During the induction period, participants received 4 cycles of nab-paclitaxel 100 mg/m^2 by intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle and carboplatin area under the curve (AUC) = 5 mg*min/mL IV on Day 1 of each 21-day cycle for 4 cycles. In the absence of clinical or radiological disease progression, participants received monotherapy with nab-paclitaxel 100 mg/m^2 by intravenous infusion on Days 1 and 8 of each 21-day cycle until disease progression or unacceptable toxicity.
Period: Induction Period
Arm/Group | Nab-Paclitaxel and Carboplatin
Started | 40
Treated Population | 40
Completed | 16
Not Completed | 24
Not completed — Death | 2
Not completed — Adverse Event | 11
Not completed — Progressive Disease (PD) | 4
Not completed — Symptomatic Deterioration | 4
Not completed — Withdrawal by Subject | 2
Not completed — Miscellaneous | 1
Period: Monotherapy Period
Arm/Group | Nab-Paclitaxel and Carboplatin
Started | 16
Completed | 0
Not Completed | 16
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Progressive Disease (PD) | 8
Not completed — Symptomatic Deterioration | 1
Not completed — Withdrawal by Subject | 2
Not completed — Study Terminated by Sponsor | 2
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Population: The treated population consisted of all participants who received at least 1 dose of investigational product (IP).
Groups:
- (Induction Period) Nab-Paclitaxel and Carboplatin: Participants received 4 cycles of nab-paclitaxel 100 mg/m^2 by intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle and carboplatin area under the curve (AUC) = 5 mg*min/mL IV on Day 1 of each 21-day cycle for 4 cycles. Participants could begin monotherapy with nab-paclitaxel in the absence of clinical or radiological disease progression.
Arm/Group | (Induction Period) Nab-Paclitaxel and Carboplatin
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated population included all participants who received at least one dose of any study drug.
  Years | 67.4 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Treated population consisted of all participants who received at least 1 dose of Investigational Product.
  Participants
    Hispanic or Latino | 3
    Not Hispanic or Latino | 37
Race [Count of Participants; unit: Participants]
  White | 37
  Black | 3
Physician Reported Eastern Cooperative Oncology Group (ECOG) Performance Status at Screening [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity) Population: The Treated population consisted of all participants who received at least 1 dose of Investigational Product.
  Participants
    0 = Fully Active | 0
    1 = Restricted in Physical Activity; Ambulatory | 0
    2 = Ambulatory and Capable of All Self-care | 40
    3 = Capable of Only Limited Self-care | 0
    4 = Completely Disabled. | 0
    5 = Dead | 0
Histology [Count of Participants; unit: Participants]
  Squamous | 15
  Non-squamous | 25
Stage of Disease at Enrollment [Count of Participants; unit: Participants] — Disease stage means how big the tumor is and how far it has spread. Disease stages range from 0 (not spread) to IV (spread throughout the body). Stage 0 - the cancer has not spread beyond the inner lining of the lung Stage I - the cancer is small and hasn't spread to the lymph nodes Stage II - the cancer has spread to some lymph nodes near the original tumor Stage III - the cancer has spread to nearby tissue or spread to far away lymph nodes Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  Participants
    Stage 0 | 0
    Stage I | 0
    Stage II | 0
    Stage IIIb | 1
    Stage IV | 39
Number of Participants with Prior Systemic Anticancer Therapies [Number; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment During the Induction Period Due to Treatment Emergent Adverse Events (TEAEs).
Description: Treatment-emergent adverse events were defined as any adverse event (AE) or serious adverse event (SAE) that occurred or worsened on or after the day of the first dose of the investigational product through 28 days after the last dose of IP. In addition, any SAE with an onset date more than 28 day after the last dose of IP that was assessed by the investigator as related to IP was considered a TEAE. A participant met the primary endpoint if: an AE was the reason for discontinuation as recorded in the electronic Case Report Form (eCRF) and the participant had no doses administered beyond Cycle 4. 95% confidence interval for the percentage was calculated using the Clopper Pearson method.
Time Frame: From date of the first dose of IP until 28 days after the last dose of IP during induction and SAEs made known to the investigator any time thereafter that are suspected of being related to IP; maximum treatment duration during induction was 3.9 months
Population: The Treated population consisted of all participants who received at least 1 dose of Investigational Product.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | (Induction Period) Nab-Paclitaxel and Carboplatin
Number analyzed (Participants) | 40
Percentage of Participants | 27 [14.60 to 43.89]

2. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment During the Induction Period (Discontinuation Rate)
Description: Discontinuation Rate was measured as Percentage of Participants who Discontinued Study Treatment During the Induction Period
Time Frame: as for outcome 1
Population: The Treated population consisted of all participants who received at least 1 dose of Investigational Product.
Measure: Number; unit: Percentage of Participants
Arm/Group | (Induction Period) Nab-Paclitaxel and Carboplatin
Number analyzed (Participants) | 40
Percentage of Participants | 60.0

3. Secondary Outcome: Dose Intensity of Nab-Paclitaxel During the Entire Study
Description: Dose intensity for nab-paclitaxel during the entire study period was (mg/m^2/week) = [cumulative dose for nab-paclitaxel in mg/m^2] / [nab-paclitaxel dosing period in weeks]
Time Frame: From Day 1 of study treatment to end of study treatment; maximum treatment duration on study was 14.1 months
Population: The treated population consisted of all participants who received at least 1 dose of Investigational Product.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Groups:
- Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel: Participants received 4 cycles of nab-paclitaxel 100 mg/m^2 by IV infusion on Days 1 and 8 of each 21-day cycle and carboplatin AUC of 5 mg*min/mL IV on Day 1 of each 21-day cycle for 4 cycles during the Induction Period. In the absence of clinical or radiological disease progression, participants moved into the monotherapy period and received nab-paclitaxel 100 mg/m^2 by IV infusion on Days 1 and 8 of each 21-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
mg/m^2/week | 52.173 (10.3066)

4. Secondary Outcome: Dose Intensity of Carboplatin During the Entire Study
Description: Dose intensity for carboplatin during the entire study period was (mg*min/mL/week) = [cumulative dose for carboplatin in mg*min/mL] / [carboplatin dosing period in weeks].
Time Frame: From Day 1 of study treatment to end of study treatment; maximum treatment duration on study was 14.1 months
Population: The treated population consisted of all participants who received at least 1 dose of investigational Product.
Measure: Mean (Standard Deviation); unit: mg*min/mL/week
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
mg*min/mL/week | 1.170 (0.4673)

5. Secondary Outcome: Percentage of Participants With Dose Reductions During the Entire Study
Description: A dose reduction occurs when the dose assigned at a visit was lower than the dose assigned at the previous visit. Dose reductions are typically caused by clinically significant laboratory abnormalities and/or treatment emergent adverse events or toxicities.
Time Frame: From day 1 of IP until 28 days after the last dose of IP; maximum treatment duration was 14.1 months during the entire study
Population: The treated population consisted of all participants who received at least 1 dose of Investigational Product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
Percentage of Participants
  nab-Paclitaxel | 32.5
  Carboplatin | 27.5

6. Secondary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time in months from day 1 of treatment to the date of disease progression based on the investigator's assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria (documented by radiological assessment) or death (any cause) on or prior to the clinical cut-off date, which ever occurred earlier. RECIST V1.1 criteria includes: - Complete Response (CR) is the disappearance of all target lesions; - Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions from baseline; - Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease (PD); - Progressive Disease is at least a 20% increase in the sum of diameters of target lesions from nadir
Time Frame: From Day 1 of study drug treatment to the date of disease progression; up to the clinical cut-off date of 24 February 2017; maximum treatment duration on study was 14.1 months
Population: The treated Population consisted of all participants who received at least 1 dose of investigational product.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
months | 4.40 [2.99 to 7.00]

7. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response or Partial Response or Continued Stable Disease (Disease Control Rate)
Description: Disease control rate was defined as the percentage of participants who had continued stable disease, complete or partial response during the course of the study, according to RECIST v1.1 guidelines, as evaluated by the investigator. RECIST V1.1 criteria includes: - Complete Response is the disappearance of all target lesions; - Partial Response is at least a 30% decrease in the sum of diameters of target lesions from baseline; - Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease; - Progressive Disease is at least a 20% increase in the sum of diameters of target lesions from nadir
Time Frame: Response assessments were evaluated every 6 weeks; up to the clinical cut-off date of 24 February 2017; maximum treatment duration on study was 14.1 months
Population: The Treated population consisted of all participants who received at least 1 dose of IP
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
Percentage of Participants | 75.0 [58.80 to 87.31]

8. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time in months between day 1 of treatment and death from any cause). Participants who were still alive as of the clinical cut-off date had their OS censored at the date of last contact or clinical cut-off, whichever was earlier. Participants who were lost to follow-up prior to the end of the study or who were withdrawn from the study were censored at the time of last contact.
Time Frame: From Day 1 of study treatment to death from any cause; up to the clinical cut-off date of 24 February 2017; maximum treatment duration on study was 14.1 months
Population: The Treated population consisted of all participants who received at least 1 dose of Investigational Product.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
months | 7.66 [4.93 to 13.17]

9. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response or Partial Response According to RECIST 1.1 Guidelines
Description: Overall tumor response is defined as the percentage of participants who achieved an objective confirmed CR (the disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions from baseline) according to RECIST V1.1 guidelines, compared with baseline where baseline was the last computed tomography (CT) scan obtained prior to or on Day 1 of study treatment.
Time Frame: Response assessments were evaluated every 2 cycles; up to the clinical cut-off date of 24 February 2017; maximum treatment duration on study was 14.1 months
Population: Participants who achieved a partial or complete response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 40
Percentage of participants | 30.0 [16.56 to 46.53]

10. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from Day 1 of study treatment to the first occurrence of response (CR or PR) according to RECIST v1.1 guidelines. RECIST V1.1 criteria includes: - A Complete Response (CR) is the disappearance of all target lesions; - A Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions from baseline
Time Frame: From Day 1 of study drug treatment to the date of first occurrence of CR or PR; up to the clinical cut-off date of 24 February 2017; maximum treatment duration on study was 14.1 months
Population: Treated Population; participants with a CR or PR
Measure: Median (Full Range); unit: Months
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 12
Months | 2.00 [1.2 to 5.7]

11. Secondary Outcome: Kaplan Meier Estimate of Duration of Response
Description: Duration of overall response was measured from the time measurement criteria were first met for CR (the disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions from baseline), whichever was first recorded, until the first date that recurrent disease or PD (at least a 20% increase in the sum of diameters of target lesions from nadir) was radiologically documented (taking as reference for PD the smallest measurements recorded on study). Median and 95% CI were estimated based on the Kaplan-Meier method.
Time Frame: as for outcome 10
Population: Participants in the Treated population with a CR or PR. Participants who were non-responders (i.e., did not achieve at least a PR) were excluded from this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Nab-Paclitaxel/Carboplatin Followed by Nab-Paclitaxel
Number analyzed (Participants) | 12
Months | 6.83 [2.10 to 11.24]

12. Secondary Outcome: Number of Participants With TEAEs During the Induction and Monotherapy Periods
Description: Treatment-emergent adverse events were defined as any adverse event or serious adverse event that occurred or worsened on or after the day of the first dose of the IP through 28 days after the last dose of IP. In addition, any SAE with an onset date more than 28 day after the last dose of IP that was assessed by the investigator as related to IP was considered a TEAE. The severity of AEs were graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild l intervention/therapy required Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death.
Time Frame: From date of the first dose of IP until 28 days after the last IP dose and SAEs made known to the investigator any time thereafter that are suspected of being related to IP; up to cutoff date of 24 Feb 2017; maximum treatment duration was 14.1 months
Population: The Treated Population consisted of all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Groups:
- Induction Period: Nab-Paclitaxel and/or Carboplatin: Participants received 4 cycles of nab-paclitaxel 100 mg/m^2 by intravenous infusion on Days 1 and 8 of each 21-day cycle and carboplatin AUC of 5 mg*min/mL IV on Day 1 of each 21-day cycle for 4 cycles.
- Monotherapy Period: Nab-Paclitaxel: Participants received 4 cycles of nab-paclitaxel 100 mg/m^2 by intravenous infusion on Days 1 and 8 of each 21-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Induction Period: Nab-Paclitaxel and/or Carboplatin | Monotherapy Period: Nab-Paclitaxel
Number analyzed (Participants) | 40 | 16
Participants
  TEAE | 40 | 14
  Serious TEAE | 20 | 4
  Grade 1/2 TEAE | 39 | 14
  Grade 3/4 TEAE | 30 | 7
  Grade 3 or Higher TEAE | 30 | 7
  Treatment-Related TEAE | 38 | 12
  Treatment-Related Serious TEAE | 13 | 0
  TEAE With Action to Reduce/Interrupt IP | 25 | 3
  Treatment-Related to Reduce or Interrupt IP | 22 | 2
  TEAE with Action Taken to Withdraw IP | 11 | 1
  Treatment-Related TEAE Action to Halt IP | 8 | 1
  TEAE with Fatal Outcome | 1 | 0
  Treatment-Related TEAE with Fatal Outcome | 0 | 0

13. Other Pre Specified Outcome: Percentage of Protocol Dose
Description: The percentage of protocol specified dose administered during the induction and monotherapy periods. Percentage of protocol dose = (dose intensity / protocol weekly dose) * 100%; the protocol weekly dose of nab-paclitaxel is 66.67 mg/m2/week; the protocol weekly dose of carboplatin was 1.67 mg*min/mL/week.
Time Frame: From Day 1 of study drug treatment to end of study drug treatment; up to clinical data cut-off date of 24 February 2017; ; maximum treatment duration was 14.1 months.
Population: The Treated Population consisted of all participants who received at least 1 dose of investigational product.
Measure: Median (Full Range); unit: Percentage of Protocol Dose
Arm/Group | Induction Period: Nab-Paclitaxel and/or Carboplatin | Monotherapy Period: Nab-Paclitaxel
Number analyzed (Participants) | 40 | 16
Percentage of Protocol Dose
  nab-Paclitaxel | 82.620 [47.11 to 101.20] | 71.185 [46.32 to 101.61]
  Carboplatin | 80.630 [19.59 to 110.31] | NA [NA to NA] — Carboplatin is not administered in the monotherapy period

ADVERSE EVENTS:
Time Frame: From date of first dose of IP until 28 days after the last dose of IP and those SAEs made known to the Investigator at any time thereafter that are suspected of being related to IP: up to the clinical cut-off date of 24 February 2017.
Description: The maximum treatment duration was 14.1 months
Groups:
- Induction: Nab-Paclitaxel/Carboplatin: Participant's received nab-paclitaxel 100 mg/m^2 intravenous infusion on Days 1 and 8 of each 21-day cycle and barboplatin AUC = 5 mg*min/mL IV on Day 1 of each 21-day cycle after completion of nab-paclitaxel infusion
- Monotherapy: Nab-Paclitaxel: Participants received nab-paclitaxel 100 mg/m^2 intravenous infusion on Days 1 and 8 of each 21-day cycle
- Follow-Up Period: Participants who discontinued IP for any reason other than lost to follow-up, entered into a follow-up period; scans were performed based on standard of care. Anti-cancer treatments were collected and participants were followed for survival every 90 days for up to 1 year. Death during follow-up is defined as any death that is more than 28 days post last dose of study drug
Arm/Group | Induction: Nab-Paclitaxel/Carboplatin | Monotherapy: Nab-Paclitaxel | Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 6/40 | 2/16 | 16/31
Serious Adverse Events (participants affected / at risk) | 20/40 | 4/16 | 0/31
Other Adverse Events (participants affected / at risk) | 40/40 | 13/16 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Nab-Paclitaxel/Carboplatin (N=40) | Monotherapy: Nab-Paclitaxel (N=16) | Follow-Up Period (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Nab-Paclitaxel/Carboplatin (N=40) | Monotherapy: Nab-Paclitaxel (N=16) | Follow-Up Period (N=31)
Anaemia (Blood and lymphatic system disorders) | 17 | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 21 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0
Asthenia (General disorders) | 9 | 1 | 0
Fatigue (General disorders) | 18 | 4 | 0
Local swelling (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 4 | 2 | 0
Pain (General disorders) | 4 | 0 | 0
Pyrexia (General disorders) | 5 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 4 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 4 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 0
Depression (Psychiatric disorders) | 4 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 3 | 2 | 0

LIMITATIONS AND CAVEATS:
Due to slower than expected enrollment, Celgene elected to end enrollment. The decision was not based on safety concerns; those enrolled continued treatment and survival follow-up until 24 February 2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene sixty days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to ninety day and must delete confidential information before submission or defer publication to permit patent applications.

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02289456/SAP_000.pdf
  • Study Protocol: ABI-007-NSCL-004ProtocolAm1RedactedFinal.12Jan 2015 (2015-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02289456/Prot_001.pdf
  • Study Protocol: ABI-007-NSCL-004.OriginalProtocolRedacted11Aug2014 (2014-08-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02289456/Prot_002.pdf